## Effect of probe material (metallic vs plastic) on periimplant probing: a randomized clinical trial

NCT ID not yet assigned

Document date: 02/11/2025







## INFORMED CONSENT OF THE STUDY PARTICIPANT

| Clinical Trial." | | |
|---|---|---|
| | | as the participant |
| | | gal representative, family member, etc. of the |
| participant, Mr./Ms | | with ID numbe |
| I DECLARE that Dr. / Dr | | , |
| (First name and two surne | ames of the investigator provid | ing the information) |
| has given me sufficient i | nformation about the study a | nd has provided me with the corresponding |
| Participant Information SI | neet. | |
| I have understood the ex | planations given to me in clea | r and simple language, and the clinician who |
| attended me has allowed | me to make all the remarks I | considered necessary and has clarified all the |
| questions I raised. | | |
| I also understand that, at | any moment and without the r | eed to give any explanation, I may revoke the |
| consent I now give and I | may withdraw from the study | whenever I wish, without having to provide |
| reasons and without any | consequences. | |
| Therefore, I state that I | am satisfied with the informa | tion received and that I give my consent to |
| participate in this study. | | |
| Signature | Signature | Signature |
| Investigator | Participant | Participant's legal representative |







INFORMED CONSENT OF THE STUDY PARTICIPANT

| VITHDRAWAL OF CONSEN | Т | |
|---|---|---|
| Mr./Ms. | | as a participant |
| with ID number | or as the legal rep | presentative, family member, etc. of the |
| participant, Mr./Ms | | with ID number |
| I DECLARE that: | | |
| Dr./ Dr | | |
| has correctly informed me | e about the study: | |
| Hospitalet de Llobregat, | day of | , 20 |
| Signature | Signature | Signature |
| Investigator | Participant | Participant's legal representative |

